CLINICAL TRIAL: NCT00544739
Title: Premature Coronary Artery Disease in Women - Risk Factors and Prognosis
Acronym: PRECADIW
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: 2 P05B 013 28
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Coronary Atherosclerosis
Keywords: Coronary Artery Disease; Premature; Female
MeSH Terms: conditions — Coronary Artery Disease; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 323 women with established coronary artery disease before 55 year of age
- 2: 347 clinically healthy, age matched women selected from the National Health Survey WOBASZ study with negative history of CVD or negative exertional chest pain.

SUMMARY:
Cardiovascular risk in women is systematically underestimated by both - society and physicians. Women younger than 50 years of age with acute coronary syndrome have 2x higher mortality compared with age-matched men. A number of common vascular-disease-related conditions are more frequent in women than in men. Women develop a more severe or different form of vascular disease then men. Variability of onset, relative risk, and the synergy of traditional and novel risk factors creates a challenge to physicians possibly resulting in suboptimal management and disregard in women presenting with angina symptoms.

During last 10 years the rise in coronary artery disease (CAD) prevalence in younger women is observed. Emerging data suggest a unique risk profile in women (hypoestrogenemia with adverse effects of a protracted dysmetabolic state). The risk factors assessment and the risk factors profiles in women that are associated with CAD may be different than in men and thus merit reassessment.

Purpose The primary objective of this study is to determine characteristics and prognosis of women with premature coronary artery disease and to evaluate the extent of atherosclerosis

DETAILED DESCRIPTION:
• Study Design Single-center, standardized, case-control study designed to assess the prevalence and significance of novel and traditional risk factors of premature coronary artery disease in women. Phase I (April 30th 2005- January 1st 2008) enrolled women with onset of symptomatic coronary artery disease before 55 years of age. The control group of 347 clinically healthy, age matched women was selected from the National Health Survey WOBASZ study (Polish Multicenter Population Study designed by Epidemiology and Cardiovascular Disease Prevention and Health Promotion Department of Institute of Cardiology) according to specifically designed questionnaire for WOBASZ study, and only subjects with negative history of CVD or negative exertional chest pain were included (Rywik S, Kupść W, Piotrowski W, et al. Wieloośrodkowe ogólnopolskie badanie stanu zdrowia ludności - projekt WOBASZ Założenia metodyczne oraz logistyka. Kardiol Pol 2005;63(supl.IV) 605:613).

Definition of premature CAD in women contained onset of coronary artery disease (myocardial infarction or coronary revascularization) before 55 years of age. Study participants are enrolled after coronary angiography and after identification and screening the age of admitted patients for acute coronary syndrome, stable angina or revascularization procedure. At the time of enrollment, participants give written informed consent for the study.

Information on demographic factors, social characterization, life style, education, anthropometric measurements, symptom characteristics and anamnesis, gynecologic history, family history on CVD and cancer, physical examination data, personal or family history of CVD, socioeconomic status, cardiovascular assessments and medication used was obtained through the use of a structured case report form questionnaire (CRF).

Additional fasting blood samples (15ml) are drawn from every individual (patients and controls) and frozen immediately at -70 for genetic study and in patients only half blood samples are centrifuged, separated, and frozen immediately at -70o after processing.

Baseline evaluation consisted of CRF data, and collection of coronary angiography, carotid ultrasonography and laboratory data.

The study protocol is approved by the Institutional Review Boards and Local Bioethics Committee.

* Follow-up All patients are contacted at 6 months after discharge from the hospital, and then every 6 months, for at least 4 years, to assess symptom status, menstrual status and occurrence of cardiovascular events (MACE) including death, nonfatal myocardial infarction, coronary revascularization, cardiac surgery and hospitalization for unstable angina.
* Study Endpoints

Primary Outcome Measures:

1. To evaluate the prevalence of atherosclerosis risk factors in women with premature CAD, including family history, social, environmental, clinical, traditional and novel risk factors, menopausal status and its association with early onset of the disease as compared to matched controls.
2. To evaluate the association of clinical factors to extent and advance of atherosclerosis
3. To evaluate predictive role of clinical factors and in particular: impaired fasting glucose, abdominal obesity, hypertension, metabolic syndrome, inflammatory markers, coexisting inflammatory and immunologic diseases on prognosis at 1 year and long-term follow-up in terms of MACE (cardiovascular death, nonfatal MI, revascularization, hospitalization due to heart failure III/IV or acute coronary syndrome)

Secondary Outcome Measures:

1. To evaluate predictive role of clinical factors and in particular: impaired fasting glucose, abdominal obesity, hypertension, metabolic syndrome, inflammatory markers, coexisting inflammatory and immunologic diseases on prognosis in terms of Vascular Events (MACE, hospitalization due to CAD progression, major arrhythmia, with ICD implantation, and stroke)
2. To evaluate predictive role of clinical factors and in particular: impaired fasting glucose, abdominal obesity, hypertension, metabolic syndrome, inflammatory markers, coexisting inflammatory and immunologic diseases on prognosis in terms of components of Vascular Events and total mortality

Endpoints assessment:

Independent endpoint classification committee comprising of 2 not involved into study procedures cardiologists will review documentation of the event and classify it.

The study may have significant implications for improvement, identification and management of female patients at risk of premature atherosclerosis providing more gender-specific data for efficacy and safety of cardiovascular medication. Better scientific recognition will result in better awareness of risk and effective prevention of coronary artery disease in young females, in optimizing the delivery of heart care to population of young women and rationale for guidelines specific for women.

ELIGIBILITY:
Inclusion Criteria:

* Patients: Consecutive women with onset of evident CAD before 55 years of age (admitted to coronary angiography because of acute coronary syndrome, stable angina or revascularization procedure)
* agreement to participate the study
* Controls : age-matched healthy women selected from participants examined between 2004-2006 in the National Health Survey - WOBASZ study with negative history of exertional chest pain, angina, hospitalization of revascularization procedures or coronary treatment.

Exclusion Criteria:

* inability to give informed consent death before discharge during the index hospitalization

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cases: Consecutive women with onset of evident CAD before 55 years of age (admitted to coronary angiography because of acute coronary syndrome, stable angina or revascularization procedure Controls: age-matched healthy women selected from participants examined between 2004-2006 in the National Health Survey - WOBASZ study with negative history of exertional chest pain, angina, hospitalization of revascularization procedures or coronary treatment
Sampling Method: Non-Probability Sample
Enrollment: 670 (Actual)
Dates: Start 2005-04; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Comparison of clinical characteristics between study group and matched controls | 1-year (short-term), 4-year (long-term)
Association of clinical factors to extent and advance of atherosclerosis | 1-year (short-term), 4-year (long-term)
Predictive role of clinical factors on prognosis in terms of MACE | 1-year (short-term), 4-year (long-term)

SECONDARY OUTCOMES:
Predictive role of clinical factors on prognosis in terms of Vascular Events | 1-year, 2-year, 3-year, 4-year
Predictive role of clinical factors on prognosis in terms of components of Vascular Events and total mortality | 1-year, 2-year, 3-year, 4-year

CONTACTS AND LOCATIONS:
Overall Officials: Barbara M Lubiszewska, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- Institute of Cardiology,, Warsaw, Poland

REFERENCES:
- [Result] Lubiszewska B, Kruk M, Broda G, Ksiezycka E, Piotrowski W, Kurjata P, Zielinski T, Ploski R. The impact of early menopause on risk of coronary artery disease (PREmature Coronary Artery Disease In Women--PRECADIW case-control study). Eur J Prev Cardiol. 2012 Feb;19(1):95-101. doi: 10.1177/1741826710394269. Epub 2011 Feb 21. PMID 21450613
- [Result] Lubiszewska B, Skora E, Kruk M, Broda G, Ksiezycka E, Kurjata P, Zielinski T, Ploski R. Prevalence of classical risk factors in Polish women with premature coronary artery disease. Kardiol Pol. 2010 Sep;68(9):1032-7. PMID 20859896